CLINICAL TRIAL: NCT03575026
Title: Partnership With the Community to Improve the Well-being of People With Mild Cognitive Impairment (MCI)/Early Dementia and Their Caregivers With Music Intervention: an Effectiveness-Implementation Cluster Randomized Clinical Hybrid Trial
Brief Title: Effectiveness-Implementation Cluster RCT to Improve Community-dwelling Early Dementia Patients by Music Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Daphne Cheung, Research Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5-ZH2P
Record Dates: First submitted 2018-04-11; First posted 2018-07-02 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Dementia
Keywords: Early dementia; Caregiver; Anxiety; Well-being
MeSH Terms: conditions — Dementia; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Subjects will receive 12-week music-with-movement intervention at home by their trained caregivers for 12 weeks, at least 3 sessions per week and 30 minutes for each session.
  Interventions: Behavioral: Music-with-movement
- Wait-list control (Placebo Comparator): Subjects will receive 12-week usual care (social activity) at home. Dose is similar to intervention arm. After the completion of 12-week usual care, subjects will receive the same music intervention as intervention arm.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Music-with-movement — Subjects will listen their preferred music and move their body actively with music
  Arms: Intervention
Behavioral: Usual care — Social activity acts as control with similar dose and intensity with intervention arm
  Arms: Wait-list control

SUMMARY:
This is a 12-week cluster randomized controlled trial utilizing music-with-movement (MWM) intervention compared with usual care to investigate the effect of MWM among subjects with early dementia or mild cognitive impairment implemented by their caregivers at home.

DETAILED DESCRIPTION:
Dementia is a neurodegenerative disorder and it can adversely affect patient's cognitive, behavioural, social and emotional functioning. Its prevalence will increase continuously because of the increase in aging population and it is predicted that around 333,000 people in Hong Kong (equivalent to 11% population aged 60 or above) will suffer from dementia in year 2039. The gradual functional decline, communication difficulties, the behavioural symptoms associated with cognitive impairment, may affect the relationships with the family members and the wellbeing. A latest Cochrane Review commented that music-based intervention may be helpful to improve emotional wellbeing and quality of life according to some limited evidences, as well as depressive symptoms, although future studies with larger sample sizes and more rigorous research design are suggested

In 2014 - 2016, our team has modified a music-with-movement intervention designed for nursing home residents with moderate dementia, into a protocol specified for caregiver-delivered home-based intervention to promote the psychosocial wellbeing of people with early dementia in Hong Kong. We found that the dyadic music-with-movement intervention yielded significant reduction on anxiety levels of people with early dementia as compared to control group. Similar, Särkämö and colleagues also found that caregiver-implemented music intervention group have reduced depression of people with early dementia and reduced caregiver burden. With the strong evidence that music intervention is useful in improving the wellbeing of people with early dementia and their family caregiver, it is essential to disseminate the culture-appropriated and validated intervention for promoting health and evaluate its effectiveness in real-practice setting by implementation research.

This research is anchored by a conceptual framework of leisure and subjective wellbeing. This framework explained that through participating in activities outside the obligated works (either paid or unpaid) that is subjectively regarded as leisure, would lead to an improvement of well-being through five psychological mechanisms, namely detachment-relaxation, autonomy, mastery, meaning and affiliation. Caregivers and care-recipients are found relaxed after participating in music intervention because they are temporary detached from the everyday caregiving chaos. Participating in an intervention designed by the participants themselves would increase their sense of autonomy and mastery. During the dyadic music intervention, the caregivers and people with MCI/early dementia would design their activities within the music-with-movement framework after instruction of music therapist that allow them to exercise their choices based on their music preference. Through the interaction in the dyadic intervention, it has been found that through participating in dyadic music intervention, people with dementia and their caregivers have improved in relationship and social inclusiveness. Caregivers would feel their competence or mastery in the skills when leading music intervention. Staff and caregivers reported that activities that address the psychological needs, provide enjoyment, value individuality, reinforce a sense of identity and belonging are meaningful to people with dementia. Therefore, we hypothesized that dyadic music-with-movement intervention would improve the subjective wellbeing of both the people with MCI/early dementia and their caregiver, if there are relevant implementation strategies to increase the ease of uptake of the intervention. For example, stress of caregivers could be relieved by successful music intervention.

When the aim is to maximize the uptake of the intervention in the real-life settings as a routine, we have to examine the influence of contextual factors on implementation. Hence, this study have three main objectives:

1. To test the effectiveness of the dyadic music-with-movement intervention on wellbeing of people with MCI/early dementia, and of their caregivers in real-life settings;
2. To conduct a process evaluation of the effectiveness-implementation study by gathering information on the implementation process; and
3. To validate and extend the applicability of "Leisure & Wellbeing" conceptual framework to the dyads.

   In this project, one of the implementation strategies to maximize the uptake of the music intervention by the dyads, is to train a team volunteers to support the caregivers and people with MCI/early dementia, which is a unique group of population. There is a general lack of knowledge and inappropriate attitude towards dementia or Alzheimer's disease worldwide. In Hong Kong, it was reported that university students majoring in medicine, nursing, occupational therapy and social work showed inadequate knowledge towards this group of patients. By providing training for volunteers to support participating dyads, it would be able to provide a better understanding on dementia and create a supportive community for dementia. Therefore, we will explore the changes in the following outcomes of the volunteers:
4. To examine the change of knowledge and attitudes towards dementia of the volunteers before and after participating in the project; and
5. To examine the change of satisfaction and motivation to volunteering before and after participating in the project.

ELIGIBILITY:
Patients with dementia/people with mild cognitive impairment

Inclusion Criteria:

* Aged 60 or above
* Cognitively impaired, defined by Global Deterioration Scale 3 or 4
* Community-dwelling
* With stable medical condition
* Able to communicate in Cantonese
* have a family caregiver who was willing to take part in the study

Exclusion Criteria:

* Suffering from any critical medical or psychiatric illnesses
* Unable to hear even using hearing aids
* Unable to sit independently for around 30 minutes
* Received music intervention within 6 months
* Participate in any clinical trial within 6 months prior to the start of study

Caregivers

Inclusion criteria:

* Primary caregiver of the PWeD
* Related to the PWeD and not a paid live-in care attendant

Exclusion criteria:

* Suffering from any critical medical or psychiatric illnesses
* Received music intervention within 6 months prior to the start of study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Changes in patients' anxiety | Baseline, immediate post-intervention (month 3)
  Rating Anxiety in Dementia (RAID), total score (range 0-54), higher indicates higher anxiety level (score>=11 indicates clinically significant anxiety)
Changes in patients' depression | Baseline, immediate post-intervention (month 3)
  Cornell scale for depression in dementia (CSDD), total score (range 0-36), higher indicates higher depression
Changes in caregivers' stress and well-being | Baseline, immediate post-intervention (month 3)
  Perceived Stress Scale 10 (PSS-10), total score (range 0-40), higher indicates higher perceived stress
Changes in caregivers' stress | Baseline, immediate post-intervention (month 3)
  Heart Rate Variability (HRV)
Changes in caregivers' well-being | Baseline, immediate post-intervention (month 3)
  Positive Aspects of Caregiving scale (PAC), total score (range 0-44), higher indicates more gain from caregiving experience
Changes in caregivers' relationship with PWD | Baseline, immediate post-intervention (month 3)
  Quality of the Caregiver-Care Recipient Relationship, 4 questions (range 0-4 each), higher score indicates better relationship between caregiver and care recipient

SECONDARY OUTCOMES:
Changes in volunteers' satisfaction from volunteering | Baseline, 3-month post-intervention (month 6)
  Volunteer Satisfaction Index (VSI), 3 sub-scores (Relationship within organization [range 0-70], Personal gain [range 0-70], Relationship with peers [range 0-28]). In any sub-score, higher mean better satisfaction in that aspect
Changes in volunteers' expectation from volunteering | Baseline, 3-month post-intervention (month 6)
  Volunteer Functions Inventory (VFI), 6 sub-scores (Protective [range 0-35], Values [range 0-35], Career [range 0-35], Social [range 0-35], Understanding [range 0-35], Enhancement [range 0-35]). In each sub-score, higher score indicates that aspect motivates more that individual to be a volunteer.
Changes in volunteers' knowledge towards dementia | Baseline, 3-month post-intervention (month 6)
  Alzheimer's Disease Knowledge Scale (ADKS), total score (range 0-24), higher indicates better knowledge towards Alzheimer's Disease
Changes in volunteers' attitude towards dementia | Baseline, 3-month post-intervention (month 6)
  Dementia Attitude Scale (DAS), total score [calculated by summation of 2 sub-scores, range 0-140] and 2 sub-scores (Comfort [range 0-70], Knowledge [range 0-70]). Higher indicates more positive attitude towards people with dementia.

OTHER OUTCOMES:
Feasibility of MWM intervention in community | 3-month post-intervention
  Interview caregivers, patients, collaborating community centre staff and supporting volunteers

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alexopoulos GS, Abrams RC, Young RC, Shamoian CA. Cornell Scale for Depression in Dementia. Biol Psychiatry. 1988 Feb 1;23(3):271-84. doi: 10.1016/0006-3223(88)90038-8. PMID 3337862
- [Background] Alexopoulos GS, Abrams RC, Young RC, Shamoian CA. Use of the Cornell scale in nondemented patients. J Am Geriatr Soc. 1988 Mar;36(3):230-6. doi: 10.1111/j.1532-5415.1988.tb01806.x. PMID 3339232
- [Background] Berntson, G. G., & Cacioppo, J. T. (2004). Heart rate variability: Stress and psychiatric conditions. In M. Malik & A. J. Camm (Eds.), Dynamic electrocardiography (pp. 57-64). Oxford, UK: Blackwell Publishing.
- [Background] Cahill S, Pierce M, Werner P, Darley A, Bobersky A. A systematic review of the public's knowledge and understanding of Alzheimer's disease and dementia. Alzheimer Dis Assoc Disord. 2015 Jul-Sep;29(3):255-75. doi: 10.1097/WAD.0000000000000102. PMID 26207322
- [Background] Carpenter BD, Balsis S, Otilingam PG, Hanson PK, Gatz M. The Alzheimer's Disease Knowledge Scale: development and psychometric properties. Gerontologist. 2009 Apr;49(2):236-47. doi: 10.1093/geront/gnp023. Epub 2009 Mar 25. PMID 19363018
- [Background] Cheung DSK, Lai CKY, Wong FKY, Leung MCP. The effects of the music-with-movement intervention on the cognitive functions of people with moderate dementia: a randomized controlled trial. Aging Ment Health. 2018 Mar;22(3):306-315. doi: 10.1080/13607863.2016.1251571. Epub 2016 Nov 7. PMID 27819483
- [Background] Clary EG, Snyder M, Ridge RD, Copeland J, Stukas AA, Haugen J, Miene P. Understanding and assessing the motivations of volunteers: a functional approach. J Pers Soc Psychol. 1998 Jun;74(6):1516-30. doi: 10.1037//0022-3514.74.6.1516. PMID 9654757
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Darragh M, Booth RJ, Koschwanez HE, Sollers J 3rd, Broadbent E. Expectation and the placebo effect in inflammatory skin reactions: a randomised-controlled trial. J Psychosom Res. 2013 May;74(5):439-43. doi: 10.1016/j.jpsychores.2012.12.010. Epub 2013 Jan 24. PMID 23597333
- [Background] Galindo-Kuhn, R., & Guzley, R. M. (2002). The volunteer satisfaction index: Construct definition, measurement, development, and validation. Journal of social service research, 28(1), 45-68.
- [Background] Harmer BJ, Orrell M. What is meaningful activity for people with dementia living in care homes? A comparison of the views of older people with dementia, staff and family carers. Aging Ment Health. 2008 Sep;12(5):548-58. doi: 10.1080/13607860802343019. PMID 18855170
- [Background] Liu H, Wang Y, Wang L. A review of non-contact, low-cost physiological information measurement based on photoplethysmographic imaging. Annu Int Conf IEEE Eng Med Biol Soc. 2012;2012:2088-91. doi: 10.1109/EMBC.2012.6346371. PMID 23366332
- [Background] Krueger, R., & Casey, M. (2015). Participants in a focus group. In R. A. Krueger & M. A. Casey (Eds.), Focus Groups: A Practical Guide for Applied Research (5th ed., pp. 77-136). Thousand Oaks, California, USA: SAGE.
- [Background] Kwok, T., Lam, K.-C., Yip, A., & Ho, F. (2011). Knowledge of dementia among undergraduates in the health and social care professions in Hong Kong. Social Work in Mental Health, 9(4), 287-301.
- [Background] Lai CK, Lai DL, Ho JS, Wong KK, Cheung DS. Interdisciplinary collaboration in the use of a music-with-movement intervention to promote the wellbeing of people with dementia and their families: Development of an evidence-based intervention protocol. Nurs Health Sci. 2016 Mar;18(1):79-84. doi: 10.1111/nhs.12238. Epub 2015 Sep 10. PMID 26354593
- [Background] Lawrence RH, Tennstedt SL, Assmann SF. Quality of the caregiver--care recipient relationship: does it offset negative consequences of caregiving for family caregivers? Psychol Aging. 1998 Mar;13(1):150-8. doi: 10.1037//0882-7974.13.1.150. PMID 9533197
- [Background] Legislative Council of the Hong Kong SAR. (2017). Care services for elderly persons with dementia. Retrieved from https://www.legco.gov.hk/research-publications/english/essentials-1617ise10-care-services-for-elderly-persons-with-dementia.htm
- [Background] Leung DY, Lam TH, Chan SS. Three versions of Perceived Stress Scale: validation in a sample of Chinese cardiac patients who smoke. BMC Public Health. 2010 Aug 25;10:513. doi: 10.1186/1471-2458-10-513. PMID 20735860
- [Background] Lin JN, Wang JJ. Psychometric evaluation of the Chinese version of the Cornell Scale for Depression in Dementia. J Nurs Res. 2008 Sep;16(3):202-10. doi: 10.1097/01.jnr.0000387307.34741.39. PMID 18792890
- [Background] Lou VW, Lau BH, Cheung KS. Positive aspects of caregiving (PAC): scale validation among Chinese dementia caregivers (CG). Arch Gerontol Geriatr. 2015 Mar-Apr;60(2):299-306. doi: 10.1016/j.archger.2014.10.019. Epub 2014 Nov 7. PMID 25488014
- [Background] McDuff D, Gontarek S, Picard R. Remote measurement of cognitive stress via heart rate variability. Annu Int Conf IEEE Eng Med Biol Soc. 2014;2014:2957-60. doi: 10.1109/EMBC.2014.6944243. PMID 25570611
- [Background] McParland P, Devine P, Innes A, Gayle V. Dementia knowledge and attitudes of the general public in Northern Ireland: an analysis of national survey data. Int Psychogeriatr. 2012 Oct;24(10):1600-13. doi: 10.1017/S1041610212000658. Epub 2012 May 17. PMID 22591515
- [Background] Montedori A, Bonacini MI, Casazza G, Luchetta ML, Duca P, Cozzolino F, Abraha I. Modified versus standard intention-to-treat reporting: are there differences in methodological quality, sponsorship, and findings in randomized trials? A cross-sectional study. Trials. 2011 Feb 28;12:58. doi: 10.1186/1745-6215-12-58. PMID 21356072
- [Background] Newman, D. B., Tay, L., & Diener, E. (2014). Leisure and subjective well-being: A model of psychological mechanisms as mediating factors. Journal of Happiness Studies, 15(3), 555-578.
- [Background] O'Connor, M. L., & McFadden, S. H. (2010). Development and psychometric validation of the Dementia Attitudes Scale. International journal of Alzheimer's disease, 2010.
- [Background] Osman SE, Tischler V, Schneider J. 'Singing for the Brain': A qualitative study exploring the health and well-being benefits of singing for people with dementia and their carers. Dementia (London). 2016 Nov;15(6):1326-1339. doi: 10.1177/1471301214556291. Epub 2014 Nov 24. PMID 25425445
- [Background] Peng RC, Zhou XL, Lin WH, Zhang YT. Extraction of heart rate variability from smartphone photoplethysmograms. Comput Math Methods Med. 2015;2015:516826. doi: 10.1155/2015/516826. Epub 2015 Jan 12. PMID 25685174
- [Background] Prince M, Bryce R, Albanese E, Wimo A, Ribeiro W, Ferri CP. The global prevalence of dementia: a systematic review and metaanalysis. Alzheimers Dement. 2013 Jan;9(1):63-75.e2. doi: 10.1016/j.jalz.2012.11.007. PMID 23305823
- [Background] Reyes del Paso GA, Langewitz W, Mulder LJ, van Roon A, Duschek S. The utility of low frequency heart rate variability as an index of sympathetic cardiac tone: a review with emphasis on a reanalysis of previous studies. Psychophysiology. 2013 May;50(5):477-87. doi: 10.1111/psyp.12027. Epub 2013 Feb 27. PMID 23445494
- [Background] Roland KP, Chappell NL. Meaningful activity for persons with dementia: family caregiver perspectives. Am J Alzheimers Dis Other Demen. 2015 Sep;30(6):559-68. doi: 10.1177/1533317515576389. Epub 2015 Mar 18. PMID 25788432
- [Background] Ryan, R. M., Patrick, H., Deci, E. L., & Williams, G. C. (2008). Facilitating health behaviour change and its maintenance: Interventions based on self-determination theory. European Health Psychologist, 10(1), 2-5.
- [Background] Sarkamo T, Tervaniemi M, Laitinen S, Numminen A, Kurki M, Johnson JK, Rantanen P. Cognitive, emotional, and social benefits of regular musical activities in early dementia: randomized controlled study. Gerontologist. 2014 Aug;54(4):634-50. doi: 10.1093/geront/gnt100. Epub 2013 Sep 5. PMID 24009169
- [Background] Shankar, K., Walker, M., Frost, D., & Orrell, M. (1999). The development of a valid and reliable scale for rating anxiety in dementia (RAID). Aging Ment Health, 3(1), 39-49.
- [Background] Sixsmith, A., & Gibson, G. (2007). Music and the wellbeing of people with dementia. Ageing & society, 27(1), 127-145.
- [Background] Tarlow, B. J., Wisniewski, S. R., Belle, S. H., Rubert, M., Ory, M. G., & Gallagher-Thompson, D. (2004). Positive aspects of caregiving: Contributions of the REACH project to the development of new measures for Alzheimer's caregiving. Research on Aging, 26(4), 429-453.
- [Background] Tarvainen MP, Niskanen JP, Lipponen JA, Ranta-Aho PO, Karjalainen PA. Kubios HRV--heart rate variability analysis software. Comput Methods Programs Biomed. 2014;113(1):210-20. doi: 10.1016/j.cmpb.2013.07.024. Epub 2013 Aug 6. PMID 24054542
- [Background] Van't Leven N, Prick AE, Groenewoud JG, Roelofs PD, de Lange J, Pot AM. Dyadic interventions for community-dwelling people with dementia and their family caregivers: a systematic review. Int Psychogeriatr. 2013 Oct;25(10):1581-603. doi: 10.1017/S1041610213000860. Epub 2013 Jul 24. PMID 23883489
- [Background] van der Steen JT, van Soest-Poortvliet MC, van der Wouden JC, Bruinsma MS, Scholten RJ, Vink AC. Music-based therapeutic interventions for people with dementia. Cochrane Database Syst Rev. 2017 May 2;5(5):CD003477. doi: 10.1002/14651858.CD003477.pub3. PMID 28462986
- [Background] Wadham O, Simpson J, Rust J, Murray C. Couples' shared experiences of dementia: a meta-synthesis of the impact upon relationships and couplehood. Aging Ment Health. 2016;20(5):463-73. doi: 10.1080/13607863.2015.1023769. Epub 2015 Mar 26. PMID 25811103
- [Background] Wong LP, Chui WH, Kwok YY. The Volunteer Satisfaction Index: A Validation Study in the Chinese Cultural Context. Soc Indic Res. 2011 Oct;104(1):19-32. doi: 10.1007/s11205-010-9715-3. Epub 2010 Sep 25. PMID 21957325
- [Background] Woo BK. Knowledge of dementia among Chinese American immigrants. Asian J Psychiatr. 2013 Aug;6(4):351-2. doi: 10.1016/j.ajp.2013.03.010. Epub 2013 May 8. No abstract available. PMID 23810148
- [Background] Wu, J., Lo, W. T., & Liu, E. S. (2009). Psychometric properties of the volunteer functions inventory with Chinese students. Journal of Community Psychology, 37(6), 769-780.
- [Background] Xia, N. (2014). Dementia literacy among nursing students in mainland China: a cross sectional study in three cities. (Master of Philosophy thesis), The University of Hong Kong, Hong Kong.
- [Background] Yu R, Chau PH, McGhee SM, Cheung WL, Chan KC, Cheung SH, Woo J. Trends in prevalence and mortality of dementia in elderly Hong Kong population: projections, disease burden, and implications for long-term care. Int J Alzheimers Dis. 2012;2012:406852. doi: 10.1155/2012/406852. Epub 2012 Oct 14. PMID 23097740
- [Derived] Cheung DSK, Ho LYW, Chan LCK, Kwok RKH, Lai CKY. A Home-Based Dyadic Music-with-Movement Intervention for People with Dementia and Caregivers: A Hybrid Type 2 Cluster-Randomized Effectiveness-Implementation Design. Clin Interv Aging. 2022 Aug 11;17:1199-1216. doi: 10.2147/CIA.S370661. eCollection 2022. PMID 35978943
- [Derived] Cheung DSK, Ho LYW, Kwok RKH, Lai DLL, Lai CKY. The effects of involvement in training and volunteering with families of people with dementia on the knowledge and attitudes of volunteers towards dementia. BMC Public Health. 2022 Feb 8;22(1):258. doi: 10.1186/s12889-022-12687-y. PMID 35135524

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/26/NCT03575026/Prot_SAP_000.pdf